CLINICAL TRIAL: NCT03683277
Title: Multicenter Open Label Phase 2 Single Arm Study of Ixazomib, Pomalidomide and Dexamethasone in Relapsed or Refractory Multiple Myeloma Characterized with Genomic Abnormalities of Adverse Adverse Prognostic
Brief Title: IPD in RRMM Characterized with Genomic Abnormalities of Adverse Prognostic
Acronym: IFM2014-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment issue, 26 patients enrolled instead of 70 initially planned
Sponsor: Intergroupe Francophone du Myelome (Network)
Collaborators: AXONAL (Unknown); Nantes University Hospital (Other); University Hospital, Grenoble (Other); Euraxi Pharma (Industry); QPS Holdings LLC (Industry); Bristol-Myers Squibb (Industry); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFM 2014-01
Record Dates: First submitted 2018-08-23; First posted 2018-09-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma; Relapsed and Refractory Multiple Myeloma; Genetic Condition
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Genetic Diseases, Inborn | interventions — ixazomib; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: All the patients will receive the same treatment until disease progression or end of study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ixazomib/Pomalidomide/Dexamethasone (Experimental): Single arm treatment organized in 2 separate phases
  Induction phase : association of Ixazomib, Pomalidomide & Dexamethasone (IPD) 21-days cycles - maximum of 17 cycles Ixazomib (tablets) 3 mg D1, D4, D8 and D11 Pomalidomide (tablets) 4mg D1 to D14 Dexamethasone (tablets) 40 mg/d D1, D8 and D15 if patient aged <75 years or Dexamethasone (tablets) 20 mg/d D1, D8 and D15 if patient aged ≥ 75 years
  Maintenance phase : association of Ixazomib and Pomalidomide (IP) 28-days cycles until disease progression Ixazomib (tablets) 4mg D1, D8 and D15 Pomalidomide (tablets) 4mg D1 to D21
  Interventions: Drug: Ixazomib/Pomalidomide/Dexamethasone

INTERVENTIONS:
Drug: Ixazomib/Pomalidomide/Dexamethasone — Treatment with association of Ixazomib, Pomalidomide and Dexamethasone (IPD)
  Induction phase : 21-days cycles - maximum of 17 cycles Ixazomib (tablets) 3 mg D1, D4, D8 and D11 Pomalidomide (tablets) 4mg D1 to D14 Dexamethasone (tablets) 40 mg/d D1, D8 and D15 if patient aged <75 years Dexamethasone (tablets) 20 mg/d D1, D8 and D15 if patient aged ≥ 75 years
  Treatment with association of Ixazomib and Pomalidomide (IP) Maintenance phase : 28-days cycles until disease progression Ixazomib (tablets) 4mg D1, D8 and D15 Pomalidomide (tablets) 4mg D1 to D21
  Other Names: Multicentric, phase 2, RRMM, refractory, relapse, myeloma

SUMMARY:
This study is a Multicenter, Open-label, Phase II study of ixazomib, plus Pomalidomide and Dexamethasone regimen (IPD) in RRMM with adverse Genomic Abnormalities.

DETAILED DESCRIPTION:
There is no escalation dose study, the maximum tolerated dose has already been determined in previous phase 1 escalation dose studies. The proposed dose of dexamethasone is considered standard. Patients will receive the IPd regimen until progression.

The hypothesis is that this IPd regimen based combination will eventually improve time to disease progression, with no additional toxicity, as compared to other available regimens, in this subgroup of patients with myeloma characterized with a very adverse prognosis.

Study design. This trial will study the efficacy and safety of IPd regimen in Relapsed and Refractory Multiple Myeloma with adverse Genomic Abnormalities until progression in 2 separate phases.

* Induction phase: 17 cycles - 21-days cycles Ixazomib 3 mg D1, D4, D8 and D11 Pomalidomide 4mg D1 to D14 Dexamethasone 40 mg/d D1, D8 and D15 if patient aged <75 years Dexamethasone 20 mg/d D1, D8 and D15 if patient aged ≥ 75 years
* Maintenance phase: until progression - 28-days cycles Ixazomib 4mg D1, D8 and D15 Pomalidomide 4mg D1 to D21
* It is not planned for the patients to receive autologous stem-cell transplantation as part of the study trial

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or older.
2. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
3. Life expectancy > 3 months.
4. Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2.
5. Presence - at diagnosis or at relapse - of one of the following adverse genomic abnormalities determined using Interphase fluorescence in situ hybridization and Single nucleotide polymorphism (FISH/SNP) techniques at a significant rate validated centrally by Pr AVET - LOISEAU:

   * deletion 17p
   * and/ or translocation (4; 14)
6. Must have an RRMM and have received a Lenalidomide line of treatment
7. Must have a Progressive Multiple Myeloma (MM) according to IMWG consensus recommendations for multiple myeloma treatment response criteria (DURIE 2007, RAJKUMAR 2011) :

   * Increase of 25% from lowest response value in any one of the following:
   * Serum M-component (absolute increase must be ≥ 0.5 g/dL),
   * Urine M-component (absolute increase must be ≥ 200 mg/24 hours),
   * Only in subjects without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC (Free Light-Chain) levels (absolute increase must be >10 mg/dL)
   * Bone marrow plasma cell percentage: the absolute percentage must be >10%
   * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
   * Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the PC (Plasma Cell) proliferative disorder
8. Must have a measurable disease as defined by the following:

   * IgG (immunoglobulin G) and IgA (immunoglobulin A) (serum M-component > 5g/l)
   * IgD (immunoglobulin D) (serum M-component > 0.5g/l)
   * Light chain (Bence Jones > 200mg/24h)
   * For MM without measurable serum or urine M protein, involved FLC ≥100 mg/l and FLC abnormal ratio.
9. Patients must meet the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
   * Total bilirubin ≤1.5 x the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   * Calculated creatinine clearance ≥ 30 mL/min MDRD (Modification of Diet in Renal Disease) formula should be used for calculating creatinine clearance values: http://mdrd.com/
10. Able to undergo antithrombotic prophylactic treatment. HBPM (low weight heparin) is preferred. In case of anti-Vitamin K Agent, INR (international normalized ratio) must be used
11. Female patients who:

    * Have been postmenopausal for at least 2 years before the screening visit, OR
    * Are surgically sterile, OR
    * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal and post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

    Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:
    * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal and post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
12. Patients agree:

    * not to share study medication with any other person and to return all unused study drugs to the investigator.
    * to abstain from donating blood while taking the study drug therapy and for one week following discontinuation of the study drug therapy.
13. Must be able to adhere to the study visit schedule and other protocol requirements including the pregnancy prevention program as detailed in section 13.4 of protocol
14. Affiliated with an appropriate social security system.

Exclusion Criteria:

1. Any other uncontrolled medical condition or comorbidity that might interfere with subject's participation.
2. Patients not having receive Lenalidomide
3. Pregnant or breast feeding females
4. Known positive for HIV or active hepatitis type B or C.
5. Patients with non-secretory MM
6. Patient with terminal renal failure that require dialysis and clearance creatinine < 30ml/min
7. Prior history of malignancies, other than multiple myeloma, unless the patients has been free of the disease for ≥ 5 years.
8. Prior local irradiation within two weeks before first dose*

   *However, an exception (that is patients allowed to remain in the treatment phase of the study) is made for radiation therapy to a pathological fracture site to enhance bone healing or to treat post-fracture pain that is refractory to narcotic analgesics because pathologic bone fractures do not by themselves fulfill a criterion for disease progression.)
9. Evidence of central nervous system (CNS) involvement
10. Unable to take corticotherapy at study entry, Ixazomib or pomalidomide
11. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
12. Ongoing Cardiac dysfunction: specify e.g. uncontrolled hypertension, MI (Myocardial Infarction) within 6 months, unstable Angina pectoris, Cardiac arrhythmia Grade 2 or higher
13. Patients planned to receive a transplantation while on IPd protocol
14. Patients who have had Ixazomib and Pomalidomide therapy as a previous line
15. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
16. Failure to have fully recovered (ie, ≤ Grade 1 toxicity) from the reversible effects of prior chemotherapy.
17. Inability or unwillingness to comply with birth control requirements
18. Unable to take antithrombotic medicines at study entry
19. Major surgery within 14 days before enrollment.
20. Systemic treatment, within 14 days before the first dose of ixazomib and Pomalidomide, with strong CYP3A (Cytochrome P450 3A) inducers (rifampicin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
21. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
22. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
23. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib and Pomalidomide including difficulty swallowing.
24. Patient has ≥ Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
25. Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not.
26. Subjects under juridical protection guardianship or tutelage measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-11-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Time to disease progression (TTP) to IPD in RRMM with adverse Genomic Abnormalities | from Cycle 1 Day 1 of Induction phase (each Cycle is 21 days) until documented disease progression or death due to disease progression, whichever came first, assessed through study completion, an average of 18 months
  Time to progression (TTP), defined as time from the first induction cycle to confirmed progressive disease (PD) per the International Myeloma Working Group criteria, or death due to progressive disease, whichever occurs first. It is noted that the events (PD or death due to PD) may include those that occur in the maintenance phase. The analysis will be performed on an Intent-To-Treat (ITT) basis and then per protocol

SECONDARY OUTCOMES:
Incidence of Serious Adverse Events and Adverse Events as assessed by CTCAE version 4.0, dose reduction or modification | after the 10th patient has completed the first cycle of treatment (Cycle is 21 days), an average of 5 months after the beginning of the study and then every 6 months through study end
  A safety Analysis will be performed after the 10th patient enrolled has finished the first cycle of treatment, without any enrollment break. The Independent Data Monitoring Committee (IDMC) will then analyzed the following:
  * Frequency of Total Serious Adverse Events (SAE)
  * Frequency of Adverse Events (AEs) Grade 3 or higher
  * Frequency of dose reductions
  * Frequency of dose discontinuations
  Data Monitoring Committee. No enrollment break is planned unless requested by the IDMC. The IDMC will analyze:
  The interim safety analysis after the10th patient enrolled has finished the first cycle of treatment.
  Safety review along study if asked by the sponsor.
Plasma concentrations of ixazomib after twice-weekly dosing in combination with Pomalidomide and Dexamethasone | from Cycle 1 Day 1 to Cycle 5 day 1 of Induction phase (each cycle is 21 days)
  Sparse Pharmacokinetics samples for the measurement of plasma concentrations of ixazomib will be collected in this study for the purposes of population PK and exposure-response analyses
Overall Response rate (ORR, Partial Response and better) to IPD | after completion of induction treatment of the last patient included, an average of 2 years after the beginning of the study and post maintenance treatment of the last patient included, an average of 3 years and half after the beginning of the study
  Post-induction and post-maintenance overall response rate (ORR) defined as the proportions of subjects who have achieved PR or better by the end of treatment per the IMWG criteria
Very Good Partial Response (VGPR) rate to IPD | after completion of induction treatment of the last patient included, an average of 2 years after the beginning of the study and post maintenance treatment of the last patient included, an average of 3 years and half after the beginning of the study
  rate of VGPR or better, defined as the proportions of subjects who have achieved PR or better by the end of induction phase per the IMWG criteria
Complete Response (CR) rate to IPD | after completion of induction treatment of the last patient included, an average of 2 years after the beginning of the study and post maintenance treatment of the last patient included, an average of 3 years and half after the beginning of the study
  CR rate defined as the proportions of subjects who have achieved CR by the end of Induction phase per IMWG criteria
Time to response and Response duration to IPD for responders | at the end of the study treatment, an average of 3 years and half after the beginning of the study
  at the end of the study, time to response and level of response to IPD for responders patients will be analyzed
Clinical benefit response rate to IPD | at the end of the study treatment, an average of 3 years and half after the beginning of the study
  Clinical Benefit rate (CBR), Minor Response (MR) and better will be analysed at the end of the study
Overall Survival (OS) to IPD | from the start of study treatment to death or the termination of the study, whichever came first, an average of 5 years
  Overall Survival (OS) rate defined as the time in months from start of treatment and death or the termination of the study, whichever came first
Progression free survival (PFS) to IPD | from the start of study treatment to disease progression, an average of 3 years and half
  Progression free survival (PFS) defined as the time in months from start of treatment and disease progression
Event Free survival (EFS) to IPD | from the start of study treatment to death or the termination of the study, whichever came first, an average of 5 years
  Event Free survival (EFS) to IPD defined as the time in months from start of treatment and disease recurrence or onset of disease symptoms

OTHER OUTCOMES:
Response rate to IPD with to genomic abnormalities in the bone marrow tumor plasma cells. | from the start of study treatment to the termination of the study, an average of 5 years
  Response rate defined as the proportions of subjects who show a PR or better from start of treatment and the termination of the study
Survival rate to IPD with to genomic abnormalities in the bone marrow tumor plasma cells. | from the start of study treatment to the termination of the study, an average of 5 years
  Survival rate defined as the proportions of subjects who are still alive at the termination of the study
Define the molecular characteristics of the 2 groups, ER and PR to IPD | from the start of study treatment to the termination of the study, an average of 5 years
  Definition of molecular characteristics assessed by performing whole exome sequencing (WES) and RNA-sequencing (RNA-seq)
Compare the molecular characteristics of the 2 groups, ER and PR to IPD | from the start of study treatment to the termination of the study, an average of 5 years
  Comparison of molecular characteristics by performing whole exome sequencing (WES) and RNA-sequencing (RNA-seq)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier LELEU, Pr, Principal Investigator — Poitiers University Hospital
Locations (28):
- France (28):
  - CHU Angers, Angers
  - CH Avignon - Centre Hospitalier H.Duffaut, Avignon
  - Centre hospitalier de la côte basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - CHU de Caen, Caen
  - Hôpital Privé Sévigné, Cesson-Sévigné
  - CHU Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - Centre hospitalier de Dunkerque, Dunkirk
  - CHU de Grenoble, Grenoble
  - Centre hospitalier départemental de Vendée, La Roche-sur-Yon
  - CHRU Hôpital Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - CHU Saint Eloi, Montpellier
  - CHRU Hôtel Dieu, Nantes
  - Hôpital de l'Archet 1, Nice
  - Hôpital Saint Louis, Paris
  - CHU Bordeaux - Hôpital Haut Leveque, Pessac
  - Centre Hospitalier de Périgueux, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHU de Reims Hôpital Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse
  - CHRU Bretonneau, Tours
  - Hôpitaux de Brabois - CHRU de Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Bobin A, Manier S, De Keizer J, Srimani JK, Hulin C, Karlin L, Caillot D, Lafon I, Mariette C, Araujo C, Arnulf B, Bareau B, Belhadj K, Benboubker L, Braun T, Calmettes C, Decaux O, Dib M, Demarquette H, Jacquet C, Sonntag C, Godet S, Jaccard A, Lenain P, Macro M, Richez-Olivier V, Tiab M, Vincent L, Zerazhi H, Petillon MO, Rollet S, Gardeney H, Durand G, Levy A, Touzeau C, Perrot A, Moreau P, Facon T, Corre J, Ragot S, Avet-Loiseau H, Leleu X. Ixazomib, pomalidomide and dexamethasone in relapsed or refractory multiple myeloma characterized with highrisk cytogenetics: the IFM 2014-01 study. Haematologica. 2025 Mar 1;110(3):758-763. doi: 10.3324/haematol.2024.285916. No abstract available. PMID 39540213
- [Background] Assouline, S., et al. Once-weekly MLN9708, an investigational proteasome inhibitor, in patients with relapsed/refractory lymphoma: results of a phase 1 dose-escalation study in 17th EHA Annual Congress. 2012. Amsterdam, the Netherlands
- [Background] Avet-Loiseau H, Attal M, Moreau P, Charbonnel C, Garban F, Hulin C, Leyvraz S, Michallet M, Yakoub-Agha I, Garderet L, Marit G, Michaux L, Voillat L, Renaud M, Grosbois B, Guillerm G, Benboubker L, Monconduit M, Thieblemont C, Casassus P, Caillot D, Stoppa AM, Sotto JJ, Wetterwald M, Dumontet C, Fuzibet JG, Azais I, Dorvaux V, Zandecki M, Bataille R, Minvielle S, Harousseau JL, Facon T, Mathiot C. Genetic abnormalities and survival in multiple myeloma: the experience of the Intergroupe Francophone du Myelome. Blood. 2007 Apr 15;109(8):3489-95. doi: 10.1182/blood-2006-08-040410. Epub 2007 Jan 5. PMID 17209057
- [Background] Avet-Loiseau H, Attal M, Campion L, Caillot D, Hulin C, Marit G, Stoppa AM, Voillat L, Wetterwald M, Pegourie B, Voog E, Tiab M, Banos A, Jaubert J, Bouscary D, Macro M, Kolb B, Traulle C, Mathiot C, Magrangeas F, Minvielle S, Facon T, Moreau P. Long-term analysis of the IFM 99 trials for myeloma: cytogenetic abnormalities [t(4;14), del(17p), 1q gains] play a major role in defining long-term survival. J Clin Oncol. 2012 Jun 1;30(16):1949-52. doi: 10.1200/JCO.2011.36.5726. Epub 2012 Apr 30. PMID 22547600
- [Background] Avet-Loiseau H, Leleu X, Roussel M, Moreau P, Guerin-Charbonnel C, Caillot D, Marit G, Benboubker L, Voillat L, Mathiot C, Kolb B, Macro M, Campion L, Wetterwald M, Stoppa AM, Hulin C, Facon T, Attal M, Minvielle S, Harousseau JL. Bortezomib plus dexamethasone induction improves outcome of patients with t(4;14) myeloma but not outcome of patients with del(17p). J Clin Oncol. 2010 Oct 20;28(30):4630-4. doi: 10.1200/JCO.2010.28.3945. Epub 2010 Jul 19. PMID 20644101
- [Background] Bergsagel PL, Mateos MV, Gutierrez NC, Rajkumar SV, San Miguel JF. Improving overall survival and overcoming adverse prognosis in the treatment of cytogenetically high-risk multiple myeloma. Blood. 2013 Feb 7;121(6):884-92. doi: 10.1182/blood-2012-05-432203. Epub 2012 Nov 19. PMID 23165477
- [Background] Chauhan D, Tian Z, Zhou B, Kuhn D, Orlowski R, Raje N, Richardson P, Anderson KC. In vitro and in vivo selective antitumor activity of a novel orally bioavailable proteasome inhibitor MLN9708 against multiple myeloma cells. Clin Cancer Res. 2011 Aug 15;17(16):5311-21. doi: 10.1158/1078-0432.CCR-11-0476. Epub 2011 Jun 30. PMID 21724551
- [Background] Chow, L.Q., et al. MLN9708, an investigational proteasome inhibitor, in patients with solid tumors; Updated phase 1 results in Head and Neck Symposium. 2012. Phoenix, AZ
- [Background] Munshi NC, Anderson KC, Bergsagel PL, Shaughnessy J, Palumbo A, Durie B, Fonseca R, Stewart AK, Harousseau JL, Dimopoulos M, Jagannath S, Hajek R, Sezer O, Kyle R, Sonneveld P, Cavo M, Rajkumar SV, San Miguel J, Crowley J, Avet-Loiseau H; International Myeloma Workshop Consensus Panel 2. Consensus recommendations for risk stratification in multiple myeloma: report of the International Myeloma Workshop Consensus Panel 2. Blood. 2011 May 5;117(18):4696-700. doi: 10.1182/blood-2010-10-300970. Epub 2011 Feb 3. PMID 21292777
- [Background] Debes-Marun CS, Dewald GW, Bryant S, Picken E, Santana-Davila R, Gonzalez-Paz N, Winkler JM, Kyle RA, Gertz MA, Witzig TE, Dispenzieri A, Lacy MQ, Rajkumar SV, Lust JA, Greipp PR, Fonseca R. Chromosome abnormalities clustering and its implications for pathogenesis and prognosis in myeloma. Leukemia. 2003 Feb;17(2):427-36. doi: 10.1038/sj.leu.2402797. PMID 12592343
- [Background] Dewald GW, Therneau T, Larson D, Lee YK, Fink S, Smoley S, Paternoster S, Adeyinka A, Ketterling R, Van Dyke DL, Fonseca R, Kyle R. Relationship of patient survival and chromosome anomalies detected in metaphase and/or interphase cells at diagnosis of myeloma. Blood. 2005 Nov 15;106(10):3553-8. doi: 10.1182/blood-2005-05-1981. Epub 2005 Jul 19. PMID 16030187
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Fonseca R, Blood E, Rue M, Harrington D, Oken MM, Kyle RA, Dewald GW, Van Ness B, Van Wier SA, Henderson KJ, Bailey RJ, Greipp PR. Clinical and biologic implications of recurrent genomic aberrations in myeloma. Blood. 2003 Jun 1;101(11):4569-75. doi: 10.1182/blood-2002-10-3017. Epub 2003 Feb 6. PMID 12576322
- [Background] Gertz MA, Lacy MQ, Dispenzieri A, Greipp PR, Litzow MR, Henderson KJ, Van Wier SA, Ahmann GJ, Fonseca R. Clinical implications of t(11;14)(q13;q32), t(4;14)(p16.3;q32), and -17p13 in myeloma patients treated with high-dose therapy. Blood. 2005 Oct 15;106(8):2837-40. doi: 10.1182/blood-2005-04-1411. Epub 2005 Jun 23. PMID 15976175
- [Background] Gupta, N., M. Saleh, and K. Venkatakrishnan. Flat-Dosing Versus BSA-Based Dosing for MLN9708, An Investigational Proteasome Inhibitor: Population Pharmacokinetic (PK) Analysis of Pooled Data From 4 Phase-1 Studies in 53rd ASH Annual Meeting and Exposition. 2011. San Diego, CA; p. abstr 1433
- [Background] Gupta, N., et al., Clinical Pharmacokinetics of Intravenous and Oral MLN9708, An Investigational Proteasome Inhibitor: An Analysis of Data From Four Phase 1 Monotherapy Studies. in 52nd ASH Annual Meeting and Exposition, 2010. 116(21): p. abstr 1813.
- [Background] Jagannath S, Richardson PG, Sonneveld P, Schuster MW, Irwin D, Stadtmauer EA, Facon T, Harousseau JL, Cowan JM, Anderson KC. Bortezomib appears to overcome the poor prognosis conferred by chromosome 13 deletion in phase 2 and 3 trials. Leukemia. 2007 Jan;21(1):151-7. doi: 10.1038/sj.leu.2404442. Epub 2006 Nov 9. PMID 17096017
- [Background] Kumar SK, Lee JH, Lahuerta JJ, Morgan G, Richardson PG, Crowley J, Haessler J, Feather J, Hoering A, Moreau P, LeLeu X, Hulin C, Klein SK, Sonneveld P, Siegel D, Blade J, Goldschmidt H, Jagannath S, Miguel JS, Orlowski R, Palumbo A, Sezer O, Rajkumar SV, Durie BG; International Myeloma Working Group. Risk of progression and survival in multiple myeloma relapsing after therapy with IMiDs and bortezomib: a multicenter international myeloma working group study. Leukemia. 2012 Jan;26(1):149-57. doi: 10.1038/leu.2011.196. Epub 2011 Jul 29. PMID 21799510
- [Background] Kumar SK, Berdeja JG, Niesvizky R, et al. A phase 1/2 study of weekly MLN9708, an investigational oral proteasome inhibitor, in combination with lenalidomide and dexamethasone in patients with previously untreated multiple myeloma (MM). Blood. 2012;120(21):332 (abstract 332).
- [Background] Kumar S, Niesvizky R, Berdeja J, Bensinger W, Zimmerman T, Berenson J, et al. Safety and Pharmacokinetics of Weekly MLN9708, an Investigational Oral Proteasome Inhibitor, Alone and in Combination. Clinical Lymphoma Myeloma and Leukemia 2013;13(Supplement 1):S154; abstr P-230
- [Background] Kumar S, Bensinger W, Reeder C, Zimmerman T, Berenson J, Liu G, et al. Weekly dosing of the investigational oral proteasome inhibitor MLN9708 in patients (pts) with relapsed/refractory multiple myeloma (MM): A phase I study. Journal of Clinical Oncology 2012 ASCO Annual Meeting Proceedings 2012:Abstract 8034.
- [Background] Kumar S, Bensinger W, Reeder C, Zimmerman T, Berenson J, Berg D, et al. Weekly Dosing of the Investigational Oral Proteasome Inhibitor MLN9708 in Patients with Relapsed and/or Refractory Multiple Myeloma: Results From a Phase 1 Dose- Escalation Study In: 53rd ASH Annual Meeting and Exposition; 2011 10-13 Dec; San Diego, CA; p. abstr 816.
- [Background] Kumar, S. et al. A Phase 1/2 Study of Weekly MLN9708, an Investigational Oral Proteasome Inhibitor, in Combination with Lenalidomide and Dexamethasone in Patients with Previously Untreated Multiple Myeloma (MM) in 54th ASH Annual Meeting and Exposition. 2012. Atlanta, Georgia.
- [Background] Leleu X, Attal M, Arnulf B, Moreau P, Traulle C, Marit G, Mathiot C, Petillon MO, Macro M, Roussel M, Pegourie B, Kolb B, Stoppa AM, Hennache B, Brechignac S, Meuleman N, Thielemans B, Garderet L, Royer B, Hulin C, Benboubker L, Decaux O, Escoffre-Barbe M, Michallet M, Caillot D, Fermand JP, Avet-Loiseau H, Facon T; Intergroupe Francophone du Myelome. Pomalidomide plus low-dose dexamethasone is active and well tolerated in bortezomib and lenalidomide-refractory multiple myeloma: Intergroupe Francophone du Myelome 2009-02. Blood. 2013 Mar 14;121(11):1968-75. doi: 10.1182/blood-2012-09-452375. Epub 2013 Jan 14. PMID 23319574
- [Background] Lonial S, Baz R, Wang M, Talpaz M, Liu G, Berg D, et al. Phase I study of twice weekly dosing of the investigational oral proteasome inhibitor MLN9708 in patients (pts) with relapsed and/or refractory multiple myeloma (MM). J Clin Oncol (ASCO Meeting Abstracts) 2012;30(15 suppl):abstr 8017.
- [Background] Merlini, G., et al. MLN9708, a Novel, Investigational Oral Proteasome Inhibitor, in Patients with Relapsed or Refractory Light-Chain Amyloidosis (AL): Results of a Phase 1 Study in 54th ASH Annual Meeting and Exposition. 2012. Atlanta, Georgia
- [Background] Moreau P, Attal M, Garban F, Hulin C, Facon T, Marit G, Michallet M, Doyen C, Leyvraz S, Mohty M, Wetterwald M, Mathiot C, Caillot D, Berthou C, Benboubker L, Garderet L, Chaleteix C, Traulle C, Fuzibet JG, Jaubert J, Lamy T, Casassus P, Dib M, Kolb B, Dorvaux V, Grosbois B, Yakoub-Agha I, Harousseau JL, Avet-Loiseau H; SAKK; IFM Group. Heterogeneity of t(4;14) in multiple myeloma. Long-term follow-up of 100 cases treated with tandem transplantation in IFM99 trials. Leukemia. 2007 Sep;21(9):2020-4. doi: 10.1038/sj.leu.2404832. Epub 2007 Jul 12. PMID 17625611
- [Background] Rajkumar SV, Harousseau JL, Durie B, Anderson KC, Dimopoulos M, Kyle R, Blade J, Richardson P, Orlowski R, Siegel D, Jagannath S, Facon T, Avet-Loiseau H, Lonial S, Palumbo A, Zonder J, Ludwig H, Vesole D, Sezer O, Munshi NC, San Miguel J; International Myeloma Workshop Consensus Panel 1. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011 May 5;117(18):4691-5. doi: 10.1182/blood-2010-10-299487. Epub 2011 Feb 3. PMID 21292775
- [Background] Rajkumar SV. Multiple myeloma: 2013 update on diagnosis, risk-stratification, and management. Am J Hematol. 2013 Mar;88(3):226-35. doi: 10.1002/ajh.23390. PMID 23440663
- [Background] Reece D, Song KW, Fu T, Roland B, Chang H, Horsman DE, Mansoor A, Chen C, Masih-Khan E, Trieu Y, Bruyere H, Stewart DA, Bahlis NJ. Influence of cytogenetics in patients with relapsed or refractory multiple myeloma treated with lenalidomide plus dexamethasone: adverse effect of deletion 17p13. Blood. 2009 Jul 16;114(3):522-5. doi: 10.1182/blood-2008-12-193458. Epub 2009 Mar 30. PMID 19332768
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Richardson PG, Siegel D, Baz R, Kelley SL, Munshi NC, Laubach J, Sullivan D, Alsina M, Schlossman R, Ghobrial IM, Doss D, Loughney N, McBride L, Bilotti E, Anand P, Nardelli L, Wear S, Larkins G, Chen M, Zaki MH, Jacques C, Anderson KC. Phase 1 study of pomalidomide MTD, safety, and efficacy in patients with refractory multiple myeloma who have received lenalidomide and bortezomib. Blood. 2013 Mar 14;121(11):1961-7. doi: 10.1182/blood-2012-08-450742. Epub 2012 Dec 14. PMID 23243282
- [Background] Richardson P, Baz R, Wang L, Jakubowiak A, Berg D, Liu G, et al. Investigational Agent MLN9708, An Oral Proteasome Inhibitor, in Patients (Pts) with Relapsed and/or Refractory Multiple Myeloma (MM): Results From the Expansion Cohorts of a Phase 1 Dose-Escalation Study In: 53rd ASH Annual Meeting and Exposition; 2011 10-13 Dec; San Diego, CA; p. abstr 301.
- [Background] Richardson, P.G., et al. MLN9708, an investigational proteasome inhibitor, in combination with lenalidomide and dexamethasone in previously untreated multiple myeloma patients (pts): Evaluation of weekly and twice-weekly dosing in 17th EHA Annual Congress. 2012. Amsterdam, the Netherlands
- [Background] San Miguel, J., et al. Oral MLN9708, an an investigational proteasome inhibitor, in combination with melphalan and prednisone in patients with previously untreated multiple myeloma: a phase 1 study in 17th EHA Annual Congress. 2012. Amsterdam, the Netherlands.
- [Background] Sonneveld P, Schmidt-Wolf IG, van der Holt B, El Jarari L, Bertsch U, Salwender H, Zweegman S, Vellenga E, Broyl A, Blau IW, Weisel KC, Wittebol S, Bos GM, Stevens-Kroef M, Scheid C, Pfreundschuh M, Hose D, Jauch A, van der Velde H, Raymakers R, Schaafsma MR, Kersten MJ, van Marwijk-Kooy M, Duehrsen U, Lindemann W, Wijermans PW, Lokhorst HM, Goldschmidt HM. Bortezomib induction and maintenance treatment in patients with newly diagnosed multiple myeloma: results of the randomized phase III HOVON-65/ GMMG-HD4 trial. J Clin Oncol. 2012 Aug 20;30(24):2946-55. doi: 10.1200/JCO.2011.39.6820. Epub 2012 Jul 16. PMID 22802322
- [Background] Stewart AK, Fonseca R. Review of molecular diagnostics in multiple myeloma. Expert Rev Mol Diagn. 2007 Jul;7(4):453-9. doi: 10.1586/14737159.7.4.453. PMID 17620051
- [Background] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763